CLINICAL TRIAL: NCT06210646
Title: Citicoline in Ischemic Stroke, a Randomized Controlled Trial
Brief Title: Citicoline in Ischemic Stroke, a Randomized Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, Dr., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2391988
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke
Keywords: citicoline; ischemic stroke; Egypt
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: We will conduct our randomized controlled trial, which will contain 2 arms: the citicoline arm, which consists of 400 patients who received 2000 mg citicoline once daily for 12 months, and the placebo arm, consisting of 400 patients who received 1000 mg citicoline once daily for 12 months; both groups will receive open-label double antiplatelet in the form of 75 mg aspirin, and 75 mg clopidogrel for three weeks, followed by a single antiplatelet in the form of 75 mg clopidogrel for the rest of our trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; in a one-to-one ratio, a specially trained and qualified nurse randomly assigned participants to receive either citicoline or a placebo. We prepared Sequentially numbered opaque sealed envelopes and 800 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 800. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrolment numbers starting from 1, which were mentioned on their files. Files with the same number as the patient enrolment number were opened, and the patients were assigned to receive drugs A or B. Drug A included citicoline 2000 mg, and Drug B included a citicoline 1000mg. The statistical analysis was performed by an independent statistician who did not know the treatment protocol of groups A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- citicoline 2000 mg arm (Active Comparator): The citicoline arm consists of 400 patients who received 2000 mg citicoline once daily for 12 months and an open-label double antiplatelet in the form of 75 mg aspirin and 75 mg clopidogrel for three weeks, followed by a single antiplatelet in the form of 75 mg clopidogrel for the rest of our trial.
  Interventions: Drug: Citicoline 2000
- citicoline 1000 mg arm (Active Comparator): The placebo arm consists of 400 patients who received citicoline 1000mg daily for 12 months and an open-label double antiplatelet in the form of 75 mg aspirin and 75 mg clopidogrel for three weeks, followed by a single antiplatelet in the form of 75 mg clopidogrel for the rest of our trial.
  Interventions: Drug: citocoline 1000

INTERVENTIONS:
Drug: Citicoline 2000 — The citicoline arm consists of 400 patients who received 2000 mg citicoline once daily for 12 months, and an open-label double antiplatelet in the form of 75 mg aspirin, and 75 mg clopidogrel for three weeks, followed by a single antiplatelet in the form of 75 mg clopidogrel for the rest of our trial.
  Other Names: group A
  Arms: citicoline 2000 mg arm
Drug: citocoline 1000 — The placebo arm consists of 400 patients who received a citicoline 1000 mg once daily for 12 months, an open-label double antiplatelet in the form of 75 mg aspirin, and 75 mg clopidogrel for three weeks, followed by a single antiplatelet in the form of 75 mg clopidogrel for the rest of our trial.
  Other Names: group B
  Arms: citicoline 1000 mg arm

SUMMARY:
Along with the current clinical trial, the efficacy and safety of a 2000 mg daily citicoline administered within 24 hours of the first-ever ischemic stroke and lasted 12 months compared to 1000 mg were assessed through MoCA, NIHSS, mRS, and possible adverse effects.

DETAILED DESCRIPTION:
The investigators conducted a single-blinded, placebo-controlled, randomized controlled trial between December 2022 and June 2024 after approval of the ethical committee of the faculty of medicine at Kafr el-Sheik University.

The investigators got written informed consent from all eligible patients or their first order of kin before randomization.

The study will comprise 2 arms citicoline arm, which consists of 400 patients who received 2000 mg citicoline once daily for 12 months, and the placebo arm, consisting of 400 patients who received 1000 mg citicoline once daily for 12 months; all the patients in the two groups received open-label double antiplatelet in the form of 75 mg aspirin. And 75 mg clopidogrel for three weeks, followed by a single antiplatelet in the form of 75 mg clopidogrel for the rest of our trial.

Study Procedures:

Every patient in our study will undergo:

Clinical workup: History, clinical assessment & NIHSS, and the Modified Rankin Scale and MoCA scale were recorded at baseline and then after 3 months, 6 months, and 12 months as a follow-up

Detection of Risk Factors & Profiles:

Echocardiography TTE: in indicated patients ECG Monitoring: daily ECG monitoring will be performed in indicated patients. 3- Carotid Duplex: carotid duplex in indicated patients.

4- ESR & Lipid Profile& liver functions: All will be tested routinely for all patients.

Imaging Follow UP Non-contrast CT brain on admission and MRI (stroke protocol; T1W, T2W, FLAIR, DWI, T2 Echo Gradient, MRA of all intra-cerebral vessels).

CT brain: Any patient with unexplained clinical deterioration at any time throughout his/her hospital stay will be urgently imaged by CT.

Primary End Point:

The primary efficacy outcome was the MoCA score after 6 months; the primary safety outcome was the rate of treatment-related adverse effects assessed by a follow-up questionnaire after 6 months.

• Secondary End Point: the secondary efficacy outcomes were: the MoCA after 12 months, mRS after 6 months, and mRS after 12 months, and the secondary safety outcome was the rate of treatment-related adverse effects assessed by a follow-up questionnaire after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male & female patients will be included
* Age more than 18 years.
* Patients must be treated within the first 24 hours of their initial stroke symptoms onset.
* Patients not eligible to receive TPA.
* Patients with a measurable focal neurological deficit (NIHSS score ≥ 4 and less than 21) lasting at least 60 minutes.This deficit must persist from the onset and up to the time of treatment without clinically significant improvement

Exclusion Criteria:

* Patients eligible for rTPA treatment.
* Patients with any type of aphasia
* Patients in coma: patients having a score of 2 or higher in the items regarding the level of consciousness in the NIHSS.
* CT or conventional MRI evidence of any structural brain disorder other than ischemic stroke.
* History of ventricular dysrhythmias, acute myocardial infarction within 72 hours before enrolment, unstable angina, decompensated congestive heart failure, or any other acute, severe, uncontrollable, or sustained cardiovascular condition that, in the Investigator's opinion, may interfere with effective participation in the study.
* Previous disorders that may confound the interpretation of the neurological scales.
* Drug addiction-related disorders.
* Pre-existing dementia, when dementia implies a disability, measured as a score of 2 or higher in the previous mRS.
* Patients under current treatment with citicoline.
* concomitant administration of other neuroprotectant drugs (such as nimodipine, vinpocetine, piracetam, cerebrolysine).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Value of Montreal Cognitive Assessment (MoCA) | 6 months
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  Its score ranges from zero to 30 points; the normal value is from 26 to 30; mild cognitive impairment ranges from 18 to 25, Moderate cognitive impairment ranges from 10 to 17, and severe cognitive impairment is below 10 points.
Rate of drug-related complications after 6 months | 6 months
  All side effects related to the drugs in our study will be reported

SECONDARY OUTCOMES:
Value of Montreal Cognitive Assessment (MoCA) | 12 months
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  Its score ranges from zero to 30 points; the normal value is from 26 to 30; mild cognitive impairment ranges from 18 to 25, Moderate cognitive impairment ranges from 10 to 17, and severe cognitive impairment is below 10 points.
Value of Modified Rankin Scale (mRS) at 6 months | 6 months
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; its value ranges from 0 to 6; the lower the score, the better the stroke outcome; favorable stroke outcome is considered with mRS value equals two or less.
Value of Modified Rankin Scale (mRS) at 12 months | 12 months
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; its value ranges from 0 to 6; the lower the score, the better the stroke outcome; favorable stroke outcome is considered with mRS value equals two or less.
Rate of drug-related complications after 12 months | 12 months
  All side effects related to the drugs in our study will be reported

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Study Director — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data that support the findings of this research will be available from the corresponding author M. Zeinhom upon reasonable request.

REFERENCES:
- [Background] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Adibhatla RM, Hatcher JF. Citicoline mechanisms and clinical efficacy in cerebral ischemia. J Neurosci Res. 2002 Oct 15;70(2):133-9. doi: 10.1002/jnr.10403. PMID 12271462
- [Result] Cho HJ, Kim YJ. Efficacy and safety of oral citicoline in acute ischemic stroke: drug surveillance study in 4,191 cases. Methods Find Exp Clin Pharmacol. 2009 Apr;31(3):171-6. doi: 10.1358/mf.2009.31.3.1364241. PMID 19536360
- [Result] Garcia-Cobos R, Frank-Garcia A, Gutierrez-Fernandez M, Diez-Tejedor E. Citicoline, use in cognitive decline: vascular and degenerative. J Neurol Sci. 2010 Dec 15;299(1-2):188-92. doi: 10.1016/j.jns.2010.08.027. Epub 2010 Sep 27. PMID 20875651